CLINICAL TRIAL: NCT02733978
Title: Non-invasive Oxygen-Ozone Therapy in the Treatment of Digital Ulcers in Egyptian Patients With Systemic Sclerosis
Brief Title: Ozone Therapy in the Treatment of Digital Ulcers in Patients With Systemic Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Hassanien, Dr., Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Assuit Ozone
Record Dates: First submitted 2016-03-25; First posted 2016-04-12 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Ulcer; Scleroderma
Keywords: Ozone oxygen; ulcer healing
MeSH Terms: conditions — Ulcer; Scleroderma, Diffuse

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ozone treated group (Experimental): Therapeutic effects will be graded into 4 levels from grade 0 (no change) to grade 3 (wound healing). The wound sizes will be measured at baseline and day 20, respectively. Tissue biopsies will be performed at baseline and day 20, expressions of VEGF, ETAR and AT1R autoantibodies proteins will be determined by immune-histochemical examinations
  Interventions: Device: the ozone generator device (Human Pro medic, German)
- non-ozone treated group (No Intervention): Therapeutic effects will be graded into 4 levels from grade 0 (no change) to grade 3 (wound healing). The wound sizes will be measured at baseline and day 20, respectively. Tissue biopsies will be performed at baseline and day 20, expressions of VEGF, ETAR and AT1R autoantibodies proteins will be determined by immune-histochemical examinations

INTERVENTIONS:
Device: the ozone generator device (Human Pro medic, German) — noninvasive oxygen-ozone treatments with 52 ug/mL ozone (total volume: 20-50 mL) in a special bag for 30 min per day for 20 days using the ozone generator device (Human Pro Medic, German)
  Arms: ozone treated group

SUMMARY:
Digital ulcers (DUs) in scleroderma result from recurrent Raynaud's phenomenon (RP) and microtrauma with high impact on quality of life, management of DUs is a great challenge for clinicians. Medical use of ozone (triatomic oxygen) was initiated in the 19th century. Ozone has multiple therapeutic effects in wound healing due to the property of releasing nascent oxygen, which has been shown to stimulate antioxidant enzymes.

DETAILED DESCRIPTION:
Digital ulcers (DUs) in scleroderma result from recurrent Raynaud's phenomenon (RP) and microtrauma with high impact on quality of life, management of DUs is a great challenge for clinicians. Medical use of ozone (triatomic oxygen) was initiated in the 19th century. Ozone has multiple therapeutic effects in wound healing due to the property of releasing nascent oxygen, which has been shown to stimulate antioxidant enzymes, we aim to assess the effects of ozone therapy on the healing in Scleroderma DUs and the expressions of vascular endothelial growth factor (VEGF), and endothelin-1 type A receptor (ETAR) and angiotensin II type 1 receptor (AT1R) autoantibodies level in the wounds after treatment.

ELIGIBILITY:
Inclusion Criteria:

* systemic sclerosis patients with DUs fulfilling ACR/EULAR criteria for diagnosis 2013

Exclusion Criteria:

* calcinosis ulcer traumatic ulcer vasculitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
scleroderma ulcer healing | 4 months
  Ulcer size measurement in cm
Pain | 4 months
  Using 10 cm scale

SECONDARY OUTCOMES:
Ulcer biopsy | 4 months
  Biopsy from the ulcer edge

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Elvis AM, Ekta JS. Ozone therapy: A clinical review. J Nat Sci Biol Med. 2011 Jan;2(1):66-70. doi: 10.4103/0976-9668.82319. PMID 22470237